CLINICAL TRIAL: NCT00573898
Title: Pharmacokinetics of Daptomycin in Patients Receiving Continuous Veno-Venous Hemodiafiltration (CVVHDF)
Brief Title: Daptomycin Study - Collection of Pharmacokinetic Samples in Patients With Renal Failure
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Heather Johnson, Pharm D, UPMC
Other Study IDs: PRO07060252
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Renal Failure
Keywords: daptomycin
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All of your biologic samples will be under the control of the principal investigator of this research project. To protect your confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. Samples will be kept in the investigator's laboratory located in Scaife Hall, room 812, 3500 Terrace Street. You may request to have your samples destroyed if you withdraw. The request must be in writing and samples collected and not already processed will be destroyed.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This will be a prospective, multicenter, open-labeled, non-comparative pharmacokinetic study conducted in 10 critically ill, anuric patients receiving CVVHDF. Enrollment will take place at 3-5 clinical sites in the United States. A study coordinator at each site will be identified and institutional specific processes (e.g., pharmacy records, etc.) will be utilized to identify patients. Full evaluation of inclusion and exclusion criteria will be conducted by each site's coordinator within 48 hours of initiation of daptomycin therapy. Subjects receiving daptomycin 6mg/kg (total body weight) once daily for a suspected/documented infection, as deemed necessary by the treating clinician will be screened for inclusion in the current study. Dialysate, ultrafiltrate, and blood flow rate utilized during the CVVHDF procedure will be determined by clinicians at discretion to optimize stability of patients.

Daptomycin samples will be obtained around the third dose in an attempt to achieve approximate steady-state concentrations. Pre- and post-filter blood samples will be collected simultaneously with dialysate and ultrafiltrate specimens at multiple time points. Protein binding will be assessed by filtration of the serum samples at the peak drug concentration time points.

DETAILED DESCRIPTION:
Enrollment will take place at 3-5 clinical sites in the United States. Full evaluation of inclusion and exclusion criteria will be conducted by each site's coordinator within 48 hours of initiation of daptomycin therapy. Subjects receiving daptomycin 6mg/kg (total body weight) once daily for a suspected/documented infection, as deemed necessary by the treating clinician will be screened for inclusion in the current study. Dialysate, ultrafiltrate, and blood flow rate utilized during the CVVHDF procedure will be determined by clinicians at discretion to optimize stability of patients.

Daptomycin samples will be obtained around the third dose in an attempt to achieve approximate steady-state concentrations. Pre- and post-filter blood samples will be collected simultaneously with dialysate and ultrafiltrate specimens at multiple time points. Protein binding will be assessed by filtration of the serum samples at the peak drug concentration time points.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted in adult critically ill patients receiving CVVHDF who are prescribed daptomycin 6mg/kg once daily as part of required medical care for suspected/documented infection, as deemed necessary by his or her treating clinician.

Exclusion Criteria:

* Daptomycin therapy will be chosen by the treating physician based on clinical indication and it is expected that risks of therapy will have already been considered; therefore, subjects are only to be excluded based on covariates that are expected to affect pharmacokinetics. Subjects will be excluded if they are:

  * less than 18 years of age
  * producing urine greater than 50 ml per 24 hours
  * have a life expectancy less than 96 hours
  * receiving CVVHDF utilizing rates or filters that are NOT otherwise considered "standard" by the enrolling site
  * receive less than 3 doses of daptomycin
  * participating in any other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving daptomycin
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2008-03; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study will be to determine the pharmacokinetic parameters of daptomycin 6mg/kg once daily in patients receiving CVVHDF, and the rate of drug clearance through the renal replacement apparatus. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heather Johnson, Pharm D, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States